CLINICAL TRIAL: NCT00902096
Title: Predictors of Cord Blood Immunoglobin E (IgE) Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Chien-Han Chen, Min-Sheng General Hospital
Other Study IDs: 2009008
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Atopy
Keywords: cord blood; IgE; prenatal; predictor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Prenatal factors: Prenatal factors to predict cord blood IgE

SUMMARY:
Background: Increased total serum IgE levels are a common characteristic of atopic diseases. Increased cord blood IgE levels, in conjunction with a family history of atopy, are associated with the development of allergic diseases in children. However, little is known about predictors of cord blood IgE levels.

Objective: The aim of our study was to identify predictors of cord blood IgE levels in an ongoing large birth cohort of infants with or without a family history of atopy.

Methods: Blood sampling of mothers was performed just before the delivery of newborns. Cord blood was also collected when the child was born. Maternal and cord blood was measured for IgE levels and cytokines. Questionnaires were administered after birth of the infant.

ELIGIBILITY:
Inclusion Criteria:

* Mothers in pregnancy 18 years of age or older, AND
* Mothers able to speak Chinese.

Exclusion Criteria:

* Infant delivered at less than 36 weeks' gestation,
* Infant with Apgar score in 5 minutes after birth < 7,
* Infant with a major congenital anomaly, OR
* Infant admitted to an intensive care unit.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: hospital and primary care clinic based study
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2009-04

PRIMARY OUTCOMES:
cord blood IgE | at birth

SECONDARY OUTCOMES:
Cord blood cytokines or other mediators | at birth

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Han Chen, MD, Principal Investigator — Min-Sheng General Hospital
Locations (1):
- Min-Sheng General Hospital, Taoyuan District, Taiwan